CLINICAL TRIAL: NCT06772623
Title: An Open-label Multi-Cohort Phase 1b/2 Study to Evaluate the Safety, Efficacy, and Optimal Dose of Telisotuzumab Adizutecan in Combination With a PD-1 Immune Checkpoint Inhibitor in Advanced or Metastatic Non-Squamous NSCLC With No Prior Treatment for Advanced Disease and No Actionable Genomic Alterations
Brief Title: Study to Evaluate Adverse Events and Efficacy of Intravenous (IV) Telisotuzumab Adizutecan in Combination With a PD-1 Immune Checkpoint Inhibitor in Adult Participants With Advanced or Metastatic Non-Squamous NSCLC With No Prior Treatment for Advanced Disease, and No Actionable Genomic Alterations
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M24-536; 2024-514465-18 (Other: EU CT)
Record Dates: First submitted 2025-01-09; First posted 2025-01-13 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Non Small Cell Lung Carcinoma
Keywords: Non Small Cell Lung Carcinoma; Pembrolizumab; Pemetrexed; Carboplatin; Cisplatin; Telisotuzumab Adizutecan; ABBV-400; ABBV-181; Budigalimab; AndroMETa-Lung-536
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — budigalimab; pembrolizumab; Carboplatin; Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Part 1: Telisotuzumab Adizutecan + Budigalimab (Experimental): Participants will receive several doses of telisotuzumab adizutecan in combination with budigalimab, as part of the 33 month study duration.
  Interventions: Drug: Telisotuzumab Adizutecan; Drug: Budigalimab
- Part 2 Arm 1: Telisotuzumab Adizutecan + Pembrolizumab (Experimental): Participants will receive telisotuzumab adizutecan dose A in combination with pembrolizumab, as part of the 33 month study duration.
  Interventions: Drug: Telisotuzumab Adizutecan; Drug: Pembrolizumab
- Part 2 Arm 2: Telisotuzumab Adizutecan + Pembrolizumab (Experimental): Participants will receive telisotuzumab adizutecan dose B in combination with pembrolizumab, as part of the 33 month study duration.
  Interventions: Drug: Telisotuzumab Adizutecan; Drug: Pembrolizumab
- Part 2: Standard of Care (Experimental): Participants will receive pembrolizumab, pemetrexed, and investigator's choice of carboplatin or cisplatin, followed by pembrolizumab and pemetrexed, as part of the 33 month study duration.
  Interventions: Drug: Pembrolizumab; Drug: Carboplatin; Drug: Pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Drug: Telisotuzumab Adizutecan — Intravenous (IV) Infusion
  Other Names: ABBV-400
  Arms: Part 1: Telisotuzumab Adizutecan + Budigalimab; Part 2 Arm 1: Telisotuzumab Adizutecan + Pembrolizumab; Part 2 Arm 2: Telisotuzumab Adizutecan + Pembrolizumab
Drug: Budigalimab — IV Infusion
  Other Names: ABBV-181
  Arms: Part 1: Telisotuzumab Adizutecan + Budigalimab
Drug: Pembrolizumab — IV Injection
  Arms: Part 2 Arm 1: Telisotuzumab Adizutecan + Pembrolizumab; Part 2 Arm 2: Telisotuzumab Adizutecan + Pembrolizumab; Part 2: Standard of Care
Drug: Pembrolizumab — IV Infusion
  Arms: Part 2: Standard of Care
Drug: Carboplatin — IV Infusion
  Arms: Part 2: Standard of Care
Drug: Pemetrexed — IV Infusion
  Arms: Part 2: Standard of Care
Drug: Cisplatin — IV Infusion
  Arms: Part 2: Standard of Care

SUMMARY:
Non small cell lung carcinoma (NSCLC) is the most frequently occurring histologic subtype of lung cancer and is the leading cause of cancer-related deaths worldwide. The purpose of this study is to assess adverse events and change in disease activity when Telisotuzumab Adizutecan (ABBV-400) is given in combination with a programmed cell death receptor 1 (PD1) immune checkpoint inhibitor to adult participants to treat NSCLC.

Telisotuzumab Adizutecan (ABBV-400) and budigalimab are investigational drugs being developed for the treatment of NSCLC. This study will be divided into two stages, with the first stage treating participants with several doses of telisotuzumab adizutecan in combination with budigalimab within the dose escalation regimen until the dose reached is tolerable and expected to be efficacious. In Stage 2 there will be 3 treatment groups. Two groups will receive pembrolizumab with different optimized doses of telisotuzumab adizutecan (to allow for the best dose to be studied in the future). One group will receive the standard of care (SOC) - pembrolizumab, pemetrexed, and investigator's choice of carboplatin or cisplatin, followed by pembrolizumab and pemetrexed. Approximately 252 adult participants with NSCLC will be enrolled in the study in 132 sites worldwide.

In the dose escalation stage participants will be treated with increasing intravenous (IV) doses of Telisotuzumab Adizutecan in combination with budigalimab until the dose of Telisotuzumab Adizutecan reached is tolerable and expected to be efficacious. In the dose optimization stage participants will be receive IV optimized doses of Telisotuzumab Adizutecan in combination with IV pembrolizumab, or IV SOC - pembrolizumab, pemetrexed, and investigator's choice of carboplatin or cisplatin, followed by pembrolizumab and pemetrexed. The study will run for a duration of approximately 33 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at an approved institution (hospital or clinic). The effect of the treatment will be frequently checked by medical assessments, blood tests, questionnaires and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically documented non-squamous (NSq) non small cell lung carcinoma (NSCLC) that is locally advanced or metastatic will be enrolled into the study.
* Must have measurable disease per response evaluation criteria in solid tumors (RECIST) v1.1.
* For Part 1, participants must have had no more than 1 systemic therapy for advanced disease including platinum-based chemotherapy or an immune checkpoint inhibitor (as monotherapy or in combination with chemotherapy), or appropriate targeted therapy for an actionable gene alteration, if applicable, for epidermal growth factor receptor (EGFR) wild-type (WT) NSq NSCLC.
* For Part 2, participants must have no prior systemic therapy for advanced disease, no known actionable genomic alteration.
* Must have documented programmed death ligand 1 (PD-L1) status.
* For Part 2, participant must have evaluable c-Met immunohistochemistry (IHC) result per central testing prior to randomization.
* Must have adequate organ function.

Exclusion Criteria:

* Known uncontrolled metastases to the central nervous system.
* History of interstitial lung disease (ILD) or pneumonitis that required treatment with systemic steroids, or any evidence of active ILD or pneumonitis on screening chest computed tomography (CT) scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Part 1: Dose-Limiting Toxicities (DLT)s of Telisotuzumab Adizutecan | Up to Approximately 84 Days
  DLT events are defined as clinically significant adverse events or abnormal laboratory values assessed as unrelated to disease progression, underlying disease, intercurrent illness, or concomitant medications.
Part 2: Objective Response (OR) as Assessed by Blinded Independent Central Review (BICR) | Up to Approximately 33 Months
  OR is defined as confirmed complete response (CR) or confirmed partial response (PR) per BICR based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Number of Participants with Adverse Events (AE)s | Up to Approximately 33 Months
  An adverse event is defined as any untoward medical occurrence in a participant or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Part 1 and Part 2: PFS as Assessed by Investigator | Up to Approximately 33 Months
  PFS is defined as the time from the participant's randomization date to the first occurrence of radiographic progression per Investigator based on RECIST v1.1 or death from any cause, whichever occurs earlier.
Part 1 and Part 2: DOR as Assessed by Investigator | Up to Approximately 33 Months
  DOR is defined as the time from the first documented CR or PR per investigator to the first occurrence of radiographic progression per the investigator on RECIST v1.1 or death from any cause, whichever occurs first. DOR is defined for participants with confirmed CR/PR.
Part 1 and Part 2: DC as Assessed by Investigator | Up to Approximately 33 Months
  DC is defined as best overall response of confirmed CR or confirmed PR, or SD for at least 11 weeks following randomization date based on RECIST v1.1, as determined by the Investigator.
Part 1 and Part 2: Overall Survival (OS) | Up to Approximately 33 Months
  OS is defined as the time from participant's randomization date (Part 2) or first dose date of study treatment (Part 1) to the event of death from any cause.
Programmed Death Ligand 1 (PD-L1) and c-Met Subgroups: OR | Up to Approximately 33 Months
  OR is defined as confirmed CR or confirmed PR based on RECIST v1.1.
PD-L1 and c-Met Subgroups: PFS | Up to Approximately 33 Months
  PFS is defined as the time from the participant's randomization date to the first occurrence of radiographic progression based on RECIST v1.1 or death from any cause, whichever occurs earlier.
PD-L1 and c-Met Subgroups: OS | Up to Approximately 33 Months
  OS is defined as the time from participant's randomization date (Part 2) or first dose date of study treatment (Part 1) to the event of death from any cause.
PD-L1 and c-Met Subgroups: DOR | Up to Approximately 33 Months
  DOR is defined as the time from the first documented CR or PR to the first occurrence of radiographic progression per RECIST v1.1 or death from any cause, whichever occurs first. DOR is defined for participants with confirmed CR/PR.
PD-L1 and c-Met Subgroups: DC | Up to Approximately 33 Months
  DC is defined as best overall response of confirmed CR or confirmed PR, or SD for at least 12 weeks following randomization date based on RECIST v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (50):
- United States (17):
  - Providence - St. Jude Medical Center /ID# 271414, Fullerton, California
  - FOMAT Medical Research - Clinica mi Salud by Focil Med /ID# 274450, Oxnard, California
  - UCLA - Santa Monica /ID# 271690, Santa Monica, California
  - University Of Colorado - Anschutz Medical Campus /ID# 269069, Aurora, Colorado
  - Rocky Mountain Cancer Centers - Lone Tree /ID# 272603, Lone Tree, Colorado
  - Mid Florida Hematology And Oncology Center /ID# 273777, Orange City, Florida
  - Hope And Healing Cancer Services /ID# 276223, Hinsdale, Illinois
  - Community Health Network /ID# 273437, Indianapolis, Indiana
  - Astera Cancer Care /ID# 271915, East Brunswick, New Jersey
  - New York Cancer and Blood Specialists - New York /ID# 272547, New York, New York
  - University Hospitals Cleveland Medical Center /ID# 271726, Cleveland, Ohio
  - The Mark H Zangmeister Center /ID# 272502, Columbus, Ohio
  - Spoknwrd Clinical Trials /ID# 273776, Easton, Pennsylvania
  - Millennium Research & Clinical Development /ID# 271717, Houston, Texas
  - Huntsman Cancer Institute /ID# 271686, Salt Lake City, Utah
  - Vista Oncology - East Olympia /ID# 275438, Olympia, Washington
  - Northwest Medical Specialties Tacoma /ID# 270469, Tacoma, Washington
- Belgium (2):
  - Groupe Sante CHC - Clinique du MontLegia /ID# 271760, Liège, Liege
  - AZ-Delta /ID# 272433, Roeselare, West-Vlaanderen
- France (3):
  - CHU Nantes - Hopital Laennec /ID# 268475, Saint-Herblain, Loire-Atlantique
  - Centre Antoine-Lacassagne /ID# 268486, Nice, Provence-Alpes-Côte d'Azur Region
  - Institut Gustave Roussy /ID# 258373, Villejuif, Val-de-Marne
- Germany (4):
  - Universitaetsklinikum Freiburg /ID# 268473, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsklinikum Frankfurt /ID# 268721, Frankfurt am Main, Hesse
  - Universitaetsklinikum Koeln /ID# 268489, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Jena /ID# 269700, Jena, Thuringia
- Italy (3):
  - Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST - IRCCS /ID# 268684, Meldola, Forlì-Cesena
  - IRCCS Istituti Fisioterapici Ospitalieri-Istituto Nazionale Tumori Regina Elena /ID# 268626, Rome, Roma
  - IRCCS AOU di Bologna Policlinico Sant Orsola Malpighi /ID# 268675, Bologna
- Japan (6):
  - NHO Nagoya Medical Center /ID# 272515, Nagoya, Aichi-ken
  - Aichi Cancer Center /ID# 271978, Nagoya, Aichi-ken
  - Yokohama Municipal Citizen's Hospital /ID# 271979, Yokohama, Kanagawa
  - Kyoto University Hospital /ID# 272312, Kyoto, Kyoto
  - Osaka Medical And Pharmaceutical University Hospital /ID# 273309, Takatsuki, Osaka
  - National Cancer Center Hospital /ID# 273192, Chuo-Ku, Tokyo
- Pan American Center for Oncology Trials /ID# 268827, Rio Piedras, Puerto Rico
- Spain (8):
  - Complejo Hospitalario Universitario A Coruña /ID# 271456, A Coruña, A Coruna
  - Hospital Universitario Marques de Valdecilla /ID# 271314, Santander, Cantabria
  - Hospital Universitario Virgen de la Victoria /ID# 271312, Málaga, Malaga
  - Hospital Universitario Virgen Macarena /ID# 271447, Seville, Sevilla
  - Hospital General Universitario de Alicante Doctor Balmis /ID# 271316, Alicante
  - Parc de Salut Mar - Hospital del Mar /ID# 271310, Barcelona
  - Hospital Clinic de Barcelona /ID# 271452, Barcelona
  - Hospital Santa Creu i Sant Pau /ID# 271311, Barcelona
- Taiwan (6):
  - Kaohsiung Chang Gung Memorial Hospital /ID# 268138, Kaohsiung City, Kaohsiung
  - Dalin Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation /ID# 268789, Chiayi City
  - National Taiwan University Cancer Center (Ntucc) /ID# 271586, Taipei
  - Taipei Veterans General Hospital /ID# 268787, Taipei
  - Tri-Service General Hospital /ID# 269211, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 268137, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-536